CLINICAL TRIAL: NCT02059798
Title: Urinary and Sexual Function Before and After Surgical Decompression of Cervical Myelopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Dong Sup Lee, Senior researcher, The Catholic University of Korea
Other Study IDs: L201402N1
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Myelopathy; Neurogenic Bladder; Erectile Dysfunction; Psychosexual Dysfunctions; Sexual Arousal Disorder
Keywords: Myelopathy
MeSH Terms: conditions — Spinal Cord Diseases; Urinary Bladder, Neurogenic; Erectile Dysfunction; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Decompression of cervical myelopathy: JOA (Japanese Orthopaedic Association) Scores for cervical myelopathy Compliance Rigidity activity unit

SUMMARY:
Hypotheses:

Decompressive surgery of cervical myelopathy will improve bladder function.

Decompressive surgery of cervical myelopathy will improve sexual function.

DETAILED DESCRIPTION:
The investigators will enroll consecutive cohort with cervical myelopathy who are scheduled to take surgical decompression of cervical spinal cord, aged between 25 and 65.

The exams for the patients include followings

* JOA (Japanese Orthopaedic Association) Scores for cervical myelopathy
* VAS (Visual Analog Scale) pain score
* IPSS (International Prostate Symptom Score) and IIEF (International Index of Erectile Function) in male patients
* FSFI (Female Sexual Function Index) and UDI (Urinary Distress Inventory) in female patients
* Bladder compliance, Detrusor leak point pressure, Peak detrusor pressure
* Rigidity activity unit of penis

ELIGIBILITY:
Inclusion Criteria:

* evidence of progression of motor or sensory nerve
* cervical myelopathy in magnetic resonance imaging

Exclusion Criteria:

* radical pelvic surgery
* pelvic irradiation
* evidence of brain damage (dementia, cerebrovascular disease)
* evidence of psychotic disorder

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having cervical myelopathy, aged between 25 and 65
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
JOA (Japanese Orthopaedic Association) Scores for cervical myelopathy | 6 months after surgery
  This score will provide patients' conditions at a glance.

SECONDARY OUTCOMES:
Bladder compliance | 6 months after surgery
  This will be provided by urodynamic study, and will show the intactness of Guarding reflex from upper spinal cord tract.

OTHER OUTCOMES:
Rigidity activity unit of penis | 6 months after surgery
  This study will be provided by nocturnal penile tumescence study and will show the intactness of psychogenic erectile pathway.
Female sexual function index | 6 months after surgery
  This will show the female patients' sexual arousal state.

CONTACTS AND LOCATIONS:
Overall Officials: Ilsup Kim, MD, PhD, Study Chair — The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, The Catholic University of Korea, Suwon, Gyeonggi-do, South Korea